CLINICAL TRIAL: NCT01768403
Title: Centralised Pan-Algerian Survey on the Undertreatment of Hypercholesterolemia
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CDZ-XXX-2012/1
Record Dates: First submitted 2013-01-14; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Hypercholesterolemia; Cardiovascular Disease; Hypertension; Diabetes; Coronary Heart Disease; Peripheral Arterial Disease
Keywords: Hypercholesterolemia; Cardiovascular disease; Hypertension; Coronary Heart disease; Peripheral Arterial disease
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases; Hypertension; Diabetes Mellitus; Coronary Disease; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood serum

SUMMARY:
Centralized Pan-Algerian Survey on the undertreatment of hypercholesterolemia. The purpose of this study is to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the Third Joint European Task Force guidelines in the survey population.

DETAILED DESCRIPTION:
Centralised Pan-Algerian Survey on the undertreatment of hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide informed consent and comply with the survey procedures.
* Subject is on lipid lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks.

Exclusion Criteria:

- Subjects who are unwilling or unable to provide informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Subject must be 19 years of age or older of either gender or race.
  * Subject must provide informed consent and comply with the survey procedures.
  * Subject is on lipid lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks
Sampling Method: Non-Probability Sample
Enrollment: 1236 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects achieving the LDL-C goals, according to the Third Joint European Task Force (TJETF) guidelines. | 24 weeks

SECONDARY OUTCOMES:
Number and percentage of subjects achieving LDL-C goals according to the TJETF guidelines. | 24 weeks
  In the following sub-populations: - Patients with / or not with metabolic syndrome (according to NCEP III definition), - Primary/secondary prevention patients
Number and percentage of subjects achieving LDL-C goals according to the NCEP ATP III/2004 updated NCEP ATP III and to the 2005 AFSSAPS guidelines | 24 weeks
  Overall and in the following sub-populations: Patients with/or without metabolic syndrome-Iary/IIary preven
Number and percentage of subjects achieving LDL-C goals according to the : TJETF / NCEP ATP III and 2004 updated NCEP ATP III guidelines. | 24 weeks
  For the following sub-populations: Demographic variables, CV risk factors & Lipid-lowering agent class
The association between achievement of LDL-C goals, according to the Third Joint European Task Force / NCEP ATP III / 2004 updated NCEP ATP III guidelines, and patient and physician variables, assessed by multivariate logistic regression models | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Habib BENNACEUR, MD, Study Chair — AstraZeneca; Nawel BOUTEKDJIRET, MD, Study Director — AstraZeneca; Yassin BOUHOUITA-GUERMECH, Professor, Principal Investigator — Cardiology department /Mustapha Bacha Hospital